CLINICAL TRIAL: NCT03196999
Title: Remote RePS: An Entirely Remote Study of an Attention Bias Modification Training "App" for Posttraumatic Stress Disorder
Brief Title: Remotely Resolving Psychological Stress (Remote RePS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17-22529
Record Dates: First submitted 2017-06-20; First posted 2017-06-23 (Actual); Last update posted 2018-12-07 (Actual); Status verified 2018-12

CONDITIONS: Post Traumatic Stress Disorder
Keywords: PTSD; Attention bias modification; Remote app-based study; Digital Health
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to either a threat attention bias modification training or a neutral bias modification training.
Who Masked: Participant
Masking Description: Participants will be blind to which condition they will be in.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Personalized Attention Bias Training (Active Comparator): Personalized version of ABM Training.
  Interventions: Behavioral: Personalized Attention Bias Training
- Neutral Attention Training Condition (Placebo Comparator): Non-active version of ABM training.
  Interventions: Behavioral: Neutral Attention Training Condition
- Non-Personalized Attention Bias Training (Active Comparator): Non-personalized version of ABM training.
  Interventions: Behavioral: Non-Personalized Attention Bias Training

INTERVENTIONS:
Behavioral: Personalized Attention Bias Training — This self-help program will aim to reduce neurobiological threat sensitivity with the ultimate goal of developing a low-cost and highly scalable self-help tool to alleviate symptoms of PTSD. The app can be used on an iOS compatible phone and involves a training program that aims to directly reduce threat sensitivity by modifying attention. The contents of the app will be personalized for each user.
  Arms: Personalized Attention Bias Training
Behavioral: Neutral Attention Training Condition — This self-help program is a placebo control program that will be used on an iOS compatible phone. The placebo will contain only neutral words.
  Arms: Neutral Attention Training Condition
Behavioral: Non-Personalized Attention Bias Training — This self-help program administered on an app will aim to reduce neurobiological threat sensitivity with the ultimate goal of a low-cost and highly scalable self-help tool to alleviate symptoms of PTSD. The app can be used on an iOS compatible phone and involves a training program that aims to directly reduce threat sensitivity by modifying attention. The contents of the app will be the same for each user.
  Arms: Non-Personalized Attention Bias Training

SUMMARY:
The investigators have developed a mobile app called Resolving Psychological Stress (REPS) for people with posttraumatic stress disorder (PTSD). The app will administer threat-related attention bias modification to individuals who score high on a PTSD checklist. This study will be administered remotely to individuals in the United States. The aims of the study are to explore feasibility, acceptability and usability of the app in an entirely remote study, as well as to explore the efficacy of the app at reducing attention bias and PTSD symptom severity.

DETAILED DESCRIPTION:
Posttraumatic stress disorder (PTSD) is a highly disabling disorder that affects approximately 8% of the population worldwide. Threat-related attention biases represent an important mechanism that may underlie PTSD symptoms. Such attention biases predict risk for PTSD following trauma exposure, and are thought to maintain some symptoms of PTSD. Research indicates that specific forms of computerized attention bias modification (ABM) training are effective in reducing attention bias for threat. We have developed a mobile app called REPS (Resolving Psychological Stress) to administer threat-related ABM training to people with symptoms of PTSD and have tested it in a laboratory-based pilot study of 22 people with elevated PTSD symptoms. Our preliminary data indicate that the app is highly acceptable to patients and that use of the app reduces attention bias for threat and PTSD symptom severity. The proposed study will expand on this prior lab-based study to test ABM training on an app entirely remotely. Our primary aim is to examine the feasibility, acceptability and usability of remotely administered app-based ABM training and to determine the efficacy of remote app-based ABM training in reducing attention bias and PTSD symptom severity. Our secondary aim is to examine whether a personalized version of ABM training results in greater attentional bias change and anxiety reduction compared to a non-personalized ABM training.

ELIGIBILITY:
Inclusion Criteria:

* Must own an iOS device compatible with the app (i.e. iPhones or iPod Touches)
* Must score at or above 33 on PTSD Checklist (PCL-5), which indicates clinically significant PTSD symptoms.

Exclusion Criteria:

* Active suicidal ideation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 528 (Actual)
Dates: Start 2017-11-30 (Actual); Primary Completion 2018-11-01 (Actual); Study Completion 2018-11-01 (Actual)

PRIMARY OUTCOMES:
Acceptability, feasibility and usability of completing attention bias modification via a mobile app. | Two weeks
  To examine a usability survey in which participants rate their experience of completing attention bias modification via a mobile app. Specifically, the questions regard the acceptability, feasibility, and usability to a completely remote, clinical population.
Reduction in post traumatic stress disorder (PTSD) symptoms | Two weeks
  To examine if remote app-based attention bias modification training compared to control neutral attention training reduces scores on the PTSD Checklist (PCL-5), an indication of PTSD symptom severity.

SECONDARY OUTCOMES:
Reduction of PTSD Checklist (PCL) score with personalized attention bias modification | Two weeks
  To examine if remote app-based personalized attention bias modification training (uses personalized stimuli in the training) compared to non-personalized attention bias modification training (uses a standard set of stimuli) reduces PTSD symptoms via the PCL.

CONTACTS AND LOCATIONS:
Overall Officials: Aoife S O'Donovan, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco, San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: Undecided